CLINICAL TRIAL: NCT01941901
Title: Calcium Electroporation for Treatment of Cutaneous Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Julie Gehl, Medical Doctor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AA1232
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Cutaneous Metastases
Keywords: Cutaneous metastases
MeSH Terms: interventions — Calcium Chloride; Electrochemotherapy; Bleomycin

STUDY DESIGN:
Intervention Model Description: Patients with cutanoues tumors of any cancer histology were included, and metastases were marked, numbered and photographed. Syringes with either calcium or bleomycin were prepared by a pharmacist, blinded for the treating clinician. After injection of study drug (calcium or bleomycin), electroporation was performed. Metastases were followed and at the 6 month follow-up response was recorded for treated metastases and the actual drug used for each metastasis was revealed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and treating doctor only knew the size of the treated tumor, and the injection volume, but not the content of the syringe (either calcium or bleomycin).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium electroporation (Experimental): The metastases will be treated with intratumoral injection of calcium chlorid followed by electrotransfer.
  It is a once-only treatment. Calcium chlorid concentration: 9mg/ml. Total dose: 0,5ml/cm3 tumor volume.
  Interventions: Drug: Calcium electroporation
- Electrochemotherapy with bleomycin (Active Comparator): The metastases will be treated with intratumoral injection of bleomycin followed by electrotransfer.
  It is a once only treatment. bleomycin concentration: 1000 IU/ml. Total dose: o,5 ml/cm3 tumor volume.
  Interventions: Drug: Electrochemotherapy with bleomycin

INTERVENTIONS:
Drug: Calcium electroporation — Intratumoral injection, once only treatment.
  Other Names: Calcium chloride.; ATC code: A02AC; EV substance code SUB12664MIG
  Arms: Calcium electroporation
Drug: Electrochemotherapy with bleomycin — Intratumoral injection, once only treatment
  Other Names: ATC code L01DC01; EV substance code SUB00844MIG
  Arms: Electrochemotherapy with bleomycin

SUMMARY:
The purpose of this study is to evaluate the effect of calcium electroporation on cutaneous metastases, and compare calcium electroporation with standard treatment: electrochemotherapy.

DETAILED DESCRIPTION:
Double-blinded phase II clinical study. We will compare the effect of calcium electroporation for the treatment of cutaneous metastases with standard treatment: electrochemotherapy with intratumoral injection of bleomycin. Separate randomisation will be performed and the lesions will be treated with either intratumoral injection of calcium or bleomycin. It is a once only treatment and the patients will be followed up for 6 months.

It is a non-inferiority study and we accept a difference in response on 15%.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histological confirmed cutaneous metastases of any histology.
* At least 1. cutaneous metastases between 0,5 to 3cm, available to electroporation.
* Patient should have been offered standard treatment.
* At least 2 weeks since chemotherapy or radiotherapy.
* Performance status >2 (ECOG).
* Life expectancy >3 months.
* platelet count > 50 mia/l.
* International Normalized Ratio (INR) <1,2.
* Men and women of reproductive age must use effective contraception during the study.
* Patient should be able to understand participants information.
* Signed, informed consent.

Exclusion Criteria:

* Previously treatment with bleomycin > 200.000 Units/m2.
* Allergy to bleomycin.
* Clinically significant coagulopathy.
* Pregnancy or lactation.
* Participation in other clinical trial involving experimental drugs or participation in a clinical trial within 4 weeks before study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Tumor response | After 6 months
  Response evaluated by "Response Evaluation Criteria in Solid Tumors" (RECIST) guidelines version 1.1.

SECONDARY OUTCOMES:
Adverse events to calcium electroporation | After 6 months
  Describe adverse events using Common Terminology for Adverse Events, version 4.0

OTHER OUTCOMES:
Compare tumor response of calcium electroporation with tumor response of electroporation. Response is evaluated by RECIST criteria. | After 6 months
  It is a non-inferiority study, and we accept a difference in response on 15%.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, Principal Investigator — Department of Oncology, Copenhagen University hospital, Herlev
Locations (1):
- Department of Oncology, Copenhagen University Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Falk H, Lambaa S, Johannesen HH, Wooler G, Venzo A, Gehl J. Electrochemotherapy and calcium electroporation inducing a systemic immune response with local and distant remission of tumors in a patient with malignant melanoma - a case report. Acta Oncol. 2017 Aug;56(8):1126-1131. doi: 10.1080/0284186X.2017.1290274. Epub 2017 Feb 22. No abstract available. PMID 28562201
- [Result] Falk H, Matthiessen LW, Wooler G, Gehl J. Calcium electroporation for treatment of cutaneous metastases; a randomized double-blinded phase II study, comparing the effect of calcium electroporation with electrochemotherapy. Acta Oncol. 2018 Mar;57(3):311-319. doi: 10.1080/0284186X.2017.1355109. Epub 2017 Aug 17. PMID 28816072